CLINICAL TRIAL: NCT03465618
Title: Imaging of Patients With Malignant Brain Tumors Using 89Zr-cRGDY Ultrasmall Silica Particle Tracers: A Phase 1 Microdosing Study
Brief Title: A First in Human Study Using 89Zr-cRGDY Ultrasmall Silica Particle Tracers for Malignant Brain Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-599
Record Dates: First submitted 2018-03-08; First posted 2018-03-14 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Brain Cancer; Pituitary Adenoma
Keywords: 89Zr-cRGDY Ultrasmall Silica Particle Tracers; Pet Scan; 17-599
MeSH Terms: conditions — Brain Neoplasms; Pituitary Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is a two-year microdosing study that will enroll up to 10 surgical or non-surgical patients harboring pituitary adenomas, high grade gliomas or metastatic brain tumors.
Who Masked: Outcomes Assessor
Masking Description: Two expert PET scan readers, who are board-certified in Nuclear Medicine, will be designated to read and evaluate PET-CT scans. Volumetric region-of-interest analysis and extraction of the mean and maximum standard uptake values (SUVs) will be provided. Both readers will initially be blinded to the patient's clinical information for scan interpretation. A second interpretation will then be performed after both readers are provided with clinical information about the primary tumor site.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- surgical patients (Experimental): Patients will be i.v. injected with approximately 5 mCi (~3.4-6.7 nanomoles) of 89Zr-DFO-cRGDY-PEG-Cy5-C' dots (specific activity range 750.0 - 1450 mCi/ µmol) and undergo the microdosing study for purposes of collecting particle tracer kinetic and dosimetry data. The patient's PET/CT Brain scans may be acquired prior to surgery. All non-surgical and some surgical patients (at the discretion of the physician) will undergo PET brain imaging.
  Interventions: Drug: 89Zr-DFO-cRGDY-PEG-Cy5-C' dots PET Imaging; Other: Blood and Urine samples
- non-surgical patients (Experimental): Before the patient's PET Brain scans patients will be i.v. injected with approximately 5 mCi (~3.4-6.7 nanomoles) of 89Zr-DFO-cRGDY-PEG-Cy5-C' dots (specific activity range 750.0 - 1450 mCi/ µmol) and undergo the microdosing study for purposes of collecting particle tracer kinetic and dosimetry data. All non-surgical and some surgical patients (at the discretion of the physician) will undergo PET brain imaging
  Interventions: Drug: 89Zr-DFO-cRGDY-PEG-Cy5-C' dots PET Imaging; Other: Blood and Urine samples

INTERVENTIONS:
Drug: 89Zr-DFO-cRGDY-PEG-Cy5-C' dots PET Imaging — A low dose spiral CT is performed first per the standard procedure. These images will be used for both attenuation correction and registration of the serial image set. The initial PET brain scan will be acquired up to about 24 hours post injection. Based upon the discretion of the physician, non-surgical patients have the possibility of a second scan and third up to about 48 hours post injection. The times per bed position may be adjusted after the first patient is imaged, and his/her scans evaluated. Additional low dose CT scans will be performed at the image session for attenuation correction and image registration. PET study may be done on a PET-MR scanner for ease.
Other: Blood and Urine samples — Venous blood and urine samples will be obtained at approximately 0.5 hours post injection at the end of each scan

SUMMARY:
The purpose of this study is to test if PET scans using 89Zr-DFO-cRGDY-PEG-Cy5-C' dot particles, can be used to take pictures of brain tumors. The investigators want to understand how the particles are distributed and removed from the body, which may help others be treated in the future. This will be the first time that 89Zr-DFO-cRGDY-PEG-Cy5-C' dot particles are being used in people. The amount of particles given in this study is very small compared to the amount that was used in mice animal studies.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed diagnosis of malignant primary brain tumor clinical and radiographic findings consistent with a pituitary adenoma, or known metastatic cancer with brain lesion presumed to be metastatic.
* Normal baseline cardiac function based upon pre-operative evaluation at the physcian's discretion
* All patients of childbearing age must use an acceptable form of birth control
* Women who are pre-menopausal must have a negative serum pregnancy test

Exclusion Criteria:

* Known pregnancy or breast-feeding Medical illness unrelated to the tumor which in the opinion of the attending physician and principal investigator will preclude administration of the tracer

  °This includes patients with uncontrolled infection, chronic renal insufficiency, myocardial infarction within the past 6 months, unstable angina, cardiac arrhythmias other than chronic atrial fibrillation and chronic active or persistent hepatitis, or New York Heart Association Classification III or IV heart disease
* More than one metastatic cancer active in the last 5 years
* Active metastatic cancer in addition to malignant primary brain tumor
* Weight greater than the 400-lb weight limit of the PET scanner
* Unmanageable claustrophobia
* Inability to lie in the scanner for 30 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
distribution within these high-grade gliomas | 2 years
  using serial PET imaging and/or correlative histologyFollowing tumor biopsy or surgical resection, histologic assessments will be performed using autoradiography to visualize the distribution of this agent within tumor tissue specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Moss, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm